CLINICAL TRIAL: NCT06752395
Title: Cryobiopsy-centered Versus Forceps Biopsy-centered Sampling for the Diagnosis of Peripheral Pulmonary Lesions - a Multicenter Prospective Randomized Controlled Trial
Brief Title: Cryobiopsy Vs. Forceps Biopsy for Peripheral Pulmonary Lesions
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: Erbe-med (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2306-027-128
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer (NSCLC)
Keywords: Bronchoscpy; Cryobiopsy; Forceps biopsy; Lung cancer; Radial probe EBUS
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Masking Description: Due to the nature of the procedures, blinding is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryobiopsy (Experimental): Cryobiopsy Group (Primary: Cryobiopsy, Auxiliary: Forceps Biopsy) In this group, cryobiopsy is performed as the primary biopsy method for sampling peripheral lung nodules. After the cryobiopsy is completed, forceps biopsy is conducted as an auxiliary method to obtain additional tissue samples.
  Interventions: Diagnostic Test: Transbronchial lung biopsy with radial probe endobronchial ultrasound (Cryobiopsy centered)
- Forceps biopsy (Experimental): Forceps Biopsy Group (Primary: Forceps Biopsy, Auxiliary: Cryobiopsy) In this group, forceps biopsy is performed as the primary biopsy method for sampling peripheral lung nodules. Following the forceps biopsy, cryobiopsy is conducted as an auxiliary method to obtain additional tissue samples.
  Interventions: Diagnostic Test: Transbronchial lung biopsy with radial probe endobronchial ultrasound (Forceps biopsy centered)

INTERVENTIONS:
Diagnostic Test: Transbronchial lung biopsy with radial probe endobronchial ultrasound (Cryobiopsy centered) — When the lung nodule is visualized by bronchoscope using RP-EBUS, cryobiopsy is performed, followed by forceps biopsy.
  Arms: Cryobiopsy
Diagnostic Test: Transbronchial lung biopsy with radial probe endobronchial ultrasound (Forceps biopsy centered) — When the lung nodule is visualized by bronchoscope using RP-EBUS, forceps biopsy is performed, followed by cryobiopsy.
  Arms: Forceps biopsy

SUMMARY:
This multicenter clinical trial evaluates the diagnostic yields of cryobiopsy and forceps biopsy for peripheral lung nodules. In the cryobiopsy group, cryobiopsy is the primary method, supplemented by forceps biopsy. Conversely, in the forceps biopsy group, forceps biopsy is the primary method, supplemented by cryobiopsy. The study also explores the complementary relationship between the two methods and examines differences in diagnostic rates based on the order in which the procedures are performed.

DETAILED DESCRIPTION:
This is a multi center, clinical trial evaluating the diagnostic yields of cryobiopsy and forceps biopsy methods used for the biopsy of peripheral lung nodules. In the cryobiopsy group, cryobiopsy is the primary method, with forceps biopsy used as an auxiliary technique, while in the forceps biopsy group, forceps biopsy is the primary method, with cryobiopsy as the auxiliary technique. The study also investigates the complementary relationship between these biopsy methods and evaluates differences in diagnostic rates based on the sequence of the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Obtained written informed consent
* Subjects having <30mm nodule on computed tomography
* Subjects without contraindication to brochoscopy

Exclusion Criteria:

* Patients with central lesions that can be visually confirmed by bronchoscopy or those with suspicious findings of cancer metastasis in the mediastinal lymph nodes, who do not require radial bronchial endoscopic ultrasound (RP-EBUS).
* Patients who cannot discontinue medications that increase bleeding risk, such as antiplatelet agents or anticoagulants.
* Patients with bleeding disorders (e.g., platelet count < 100,000/mm³).
* Patients with severe comorbidities (e.g., serious respiratory or cardiovascular diseases) that make bronchoscopy unsafe.
* Patients with hypersensitivity or allergies to drugs commonly used in endoscopic procedures, including lidocaine, midazolam, fentanyl, or flumazenil.
* Pregnant or breastfeeding patients.
* Patients with confirmed lung cancer undergoing rebiopsy for genetic testing or other purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The overall cumulative diagnostic yield | through study completion, an average of 1 year
  Pathologic diagnostic yield of primary method and overall procedures

SECONDARY OUTCOMES:
Diagnosis Rate According to Lesion Size | through study completion, an average of 1 year
  This outcome measures the diagnostic success rate based on the size of the peripheral lung nodule. Lesions are categorized by size (e.g., <20 mm, 20 mm-30mm) to determine whether lesion size affects the accuracy and success of the biopsy method.
Diagnosis Rate According to Malignant and Benign Disease Classification | through study completion, an average of 1 year
  This measures the diagnostic yield of cryobiopsy and forceps biopsy by differentiating between malignant and benign lesions. The diagnostic rate is compared between cases of cancerous and non-cancerous nodules to assess the performance of the biopsy methods in each category.
Diagnosis Rate According to Bronchus Sign | through study completion, an average of 1 year
  The bronchus sign refers to whether or not the lesion is connected to a bronchus, as seen on imaging. This outcome evaluates whether the presence or absence of a bronchus sign impacts the diagnostic success of the biopsies.
Diagnosis Rate According to Image Classification Detected by Radial Bronchial Endoscopic Ultrasound (RP-EBUS) | through study completion, an average of 1 year
  This outcome assesses the diagnostic rate based on the characteristics of the lesion as identified by RP-EBUS imaging (e.g., solid, partially solid, or ground-glass opacities). The study evaluates whether different imaging characteristics influence the biopsy's diagnostic accuracy.
Complication Rate | through study completion, an average of 1 year
  This outcome measures the incidence of complications (e.g., bleeding, pneumothorax) that occur during or after the biopsy procedure. The complication rates are compared between the two biopsy methods to evaluate their safety profiles.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon

IPD SHARING:
Plan to Share IPD: No